CLINICAL TRIAL: NCT01164722
Title: A Randomized Clinical Trial of Infrared Coagulator (IRC) Ablation Versus Expectant Management of Intra-Anal High Grade Intraepithelial Neoplasia (HGAIN) in HIV-infected Adults
Brief Title: Infrared Coagulator Ablation or Observation in Preventing Anal Cancer in HIV-Positive Patients With Anal Neoplasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry); University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AMC-076; U01CA121947 (NIH); AMC-076 (Other: AMC)
Record Dates: First submitted 2010-07-16; First posted 2010-07-19 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Anal Cancer; Neoplasm of Uncertain Malignant Potential; Nonneoplastic Condition; Precancerous Condition
Keywords: anal cancer; HIV infection; human papilloma virus infection; neoplasm of uncertain malignant potential; high-grade squamous intraepithelial lesion
MeSH Terms: conditions — Anus Neoplasms; Precancerous Conditions; HIV Infections; Papillomavirus Infections; Squamous Intraepithelial Lesions | interventions — Watchful Waiting; Light Coagulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: Infrared coagulator treatment (Experimental): Infrared photocoagulation therapy. The infrared coagulator (IRC) contact tip is placed in direct contact with lesion under high-resolution anoscopy (HRA) guidance. Patients then undergo IRC ablation for 1.5 second pulses. IRC ablation is reapplied until the level of submucosal vessels are reached.
  Interventions: Device: infrared photocoagulation therapy
- Arm II: Expectant management (Active Comparator): Patients receive standard of care and undergo clinical observation. After 12 months, patients may receive IRC ablation to all anal intraepithelial neoplasia lesions despite of their size.
  Interventions: Other: clinical observation

INTERVENTIONS:
Other: clinical observation — Patients undergo observation
  Arms: Arm II: Expectant management
Device: infrared photocoagulation therapy — Anal infrared coagulator ablation
  Other Names: Redfield Infrared Coagulator; Redfield IRC
  Arms: Arm I: Infrared coagulator treatment

SUMMARY:
RATIONALE: Infrared coagulator ablation may be effective in preventing the development of anal cancer in patients with anal neoplasia

PURPOSE: This randomized phase III trial is studying infrared coagulator ablation to see how well it works compared to observation in preventing anal cancer in HIV-positive patients with anal neoplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the complete response rate at 3 months and 1 year in HIV-seropositive patients with high-grade anal intraepithelial neoplasia (HGAIN) treated with infrared coagulator (IRC) ablation versus observation.

Secondary

* Determine the tolerability and safety of IRC ablation versus observation in these patients.
* Compare the proportion of patients with HGAIN at 1 year.
* Evaluate the response and recurrence rates at 1 year of individual lesions in patients treated with this regimen vs observation.
* Determine the incidence of metachronous lesions in these patients.
* Compare the response and recurrence rates at 2 years of individual lesions in patients under observation who subsequently received IRC ablation with the response and recurrence rates at 1 year in patients initially treated with IRC.

OUTLINE: This is a multicenter study. Patients are stratified according to site. Patients are randomized to 1 of 2 arms.

* Arm I: Infrared coagulator (IRC) contact tip is placed in direct contact with lesion under high-resolution anoscopy (HRA) guidance for 1.5 seconds. IRC ablation is reapplied until the level of submucosal vessels are reached.

  * One week after each IRC ablation, patients complete a questionnaire regarding pain, bleeding, and other complaints.
* Arm II: Patients receive standard of care and undergo observation. After 12 months, patients may receive IRC ablation to all anal intraepithelial neoplasia lesions.

NOTE: Patients may receive a maximum of 6 IRC treatments while on study (3 per year).

Patients undergo a physical exam, digital rectal exam, anal cytology, and HRA at baseline and periodically during study.

After completion of study therapy, patients are followed up periodically for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of high-grade anal intraepithelial neoplasia (AIN) meeting the following:

  * AIN2 and/or AIN3 confirmed by biopsy ≥ 2 weeks to ≤ 60 days before enrollment
  * 1-3 lesions with each lesion ≤ 15 mm in diameter
  * At least one high-grade AIN lesion is still visible at study entry
* HIV-infection documented by federally approved, licensed HIV-test in conjunction with screening test (e.g., ELISA, western blot, or other test)

  * HIV-infection, based on prior ELISA and western blot assays, recorded and documented by another physician, allowed provided patient undergoes an approved antibody test to confirm diagnosis
  * Patients on concurrent anti-retroviral therapy with a history of HIV-positivity based on an approved antibody test allowed
  * Detectable plasma HIV-1 RNA also allowed
* No perianal AIN, perianal condyloma, or lower vulvar intraepithelial neoplasia or condyloma requiring treatment

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Life expectancy ≥ 2 years
* CD4 count ≥ 200/mm³
* ANC > 750/mm³
* Platelet count ≥ 75,000/mm³
* Hemoglobin ≥ 9.0 g/dL
* INR and aPTT normal
* Negative pregnancy test
* Fertile patients must use effective contraception
* Female patients must have undergone cervical pap smear (if having a cervix) and gynecologic evaluation within the past 12 months
* Must be capable of complying with the requirements of this protocol
* Concurrent HPV-related disease allowed
* No history of anal cancer
* No acute infection or other serious medical illness requiring treatment within the past 14 days

  * Fungal infection of the skin or a sexually transmitted disease requiring treatment allowed
* No concurrent malignancy requiring systemic therapy

  * Kaposi sarcoma limited to the skin allowed

PRIOR CONCURRENT THERAPY:

* No prior infrared coagulator (IRC) ablation for high-grade anal intraepithelial neoplasia (HGAIN)

  * Prior HGAIN treated by any means other than IRC within the past 2 months allowed
* At least 5 days since prior coumadin or clopidogrel and ≥ 7 days after study therapy before receiving coumadin or clopidogrel again
* No concurrent anticoagulant therapy other than aspirin or NSAIDs
* More than 3 months since prior and concurrent systemic corticosteroids, cytokines, or immunomodulatory therapy (e.g., interferons) or local imiquimod
* No concurrent systemic therapy

Min Age: 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-04; Primary Completion 2015-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen E. Goldstone, MD, Principal Investigator — Laser Surgery Care
Locations (7):
- United States (7):
  - UCLA Clinical AIDS Research and Education (CARE) Center, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Laser Surgery Care, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Benaroya Research Institute at Virginia Mason Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goldstone SE, Lensing SY, Stier EA, Darragh T, Lee JY, van Zante A, Jay N, Berry-Lawhorn JM, Cranston RD, Mitsuyasu R, Aboulafia D, Palefsky JM, Wilkin T. A Randomized Clinical Trial of Infrared Coagulation Ablation Versus Active Monitoring of Intra-anal High-grade Dysplasia in Adults With Human Immunodeficiency Virus Infection: An AIDS Malignancy Consortium Trial. Clin Infect Dis. 2019 Mar 19;68(7):1204-1212. doi: 10.1093/cid/ciy615. PMID 30060087

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I: Infrared Coagulator Treatment | Arm II: Expectant Management
Started | 60 | 60
Completed | 42 | 45
Not Completed | 18 | 15
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Lost to Follow-up | 3 | 6
Not completed — met protocol criteria for non-treatment | 11 | 1
Not completed — enrolled on other study, concomitant med | 1 | 3

BASELINE CHARACTERISTICS:
Population: Enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I: Infrared Coagulator Treatment | Arm II: Expectant Management | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (9.0) | 49.0 (9.6) | 49.8 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 58 | 54 | 112
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 16 | 22
  Not Hispanic or Latino | 53 | 44 | 97
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 9 | 13 | 22
  White | 46 | 46 | 92
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Through 1 Year
Description: No detection of high grade anal intraepithelial neoplasia (HGAIN) from treatment through one year. Detection of HGAIN was based on local pathology reports.
Time Frame: 1 year post treatment
Population: All study participants who were randomized and attended the baseline visit.
Measure: Number; unit: participants
Arm/Group | Arm I: Infrared Coagulator Treatment | Arm II: Expectant Management
Number analyzed (Participants) | 60 | 60
participants | 38 | 16

2. Secondary Outcome: Tolerability and Safety of Infrared Coagulator Ablation
Description: Number of patients who experienced a serious adverse events
Time Frame: All study visits through year 2
Measure: Number; unit: participants
Arm/Group | Arm I: Infrared Coagulator Treatment | Arm II: Expectant Management
Number analyzed (Participants) | 60 | 60
participants | 8 | 6

3. Secondary Outcome: Proportion of Patients With High-grade Anal Intraepithelial Neoplasia at 1 Year
Description: Number of patients who had high grade anal intraepithelial neoplasia at one year.
Time Frame: 1 year on study
Population: Patients who had an evaluable biopsy within one year after randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I: Infrared Coagulator Treatment | Arm II: Expectant Management
Number analyzed (Participants) | 55 | 57
Participants | 15 | 40

4. Secondary Outcome: Recurrence Rate at 1 Year
Time Frame: 1 year on study
Population: Patients who were treated with IRC, no data were collected on patients on the expectant management arm
Measure: Number; unit: Percentage of lesions that recurred
Arm/Group | Arm I: Infrared Coagulator Treatment | Arm II: Expectant Management
Number analyzed (Participants) | 60 | 0
Percentage of lesions that recurred | 37 |

5. Secondary Outcome: Incidence of Metachronous Lesions
Description: Number of patients with one or more metachronous lesions
Time Frame: one year on study
Population: Patents with any biopsy from randomization to one year
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I: Infrared Coagulator Treatment | Arm II: Expectant Management
Number analyzed (Participants) | 58 | 55
Participants | 26 | 15

ADVERSE EVENTS:
Time Frame: Study duration - maximum is 24 months
Arm/Group | Arm I: Infrared Coagulator Treatment | Arm II: Expectant Management
Serious Adverse Events (participants affected / at risk) | 8/60 | 6/60
Other Adverse Events (participants affected / at risk) | 54/60 | 41/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I: Infrared Coagulator Treatment (N=60) | Arm II: Expectant Management (N=60)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Aortic Valve Disease (Cardiac disorders) | 0 | 1
Cardiac Disorders, other (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0
Retinal vacular disorder (Eye disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Infections, other (Infections and infestations) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Intraoperative musculoskeletal injury (Injury, poisoning and procedural complications) | 0 | 1
Neoplasms, unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Renal calculi (Renal and urinary disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I: Infrared Coagulator Treatment (N=60) | Arm II: Expectant Management (N=60)
Anal hemorrhage (Gastrointestinal disorders) | 4 | 6
Anal pain (Gastrointestinal disorders) | 49 | 30
Anal ulcer (Gastrointestinal disorders) | 14 | 4
Diarrhea (Gastrointestinal disorders) | 6 | 4
Hemorrhoids (Gastrointestinal disorders) | 5 | 1
Flu-like symptoms (General disorders) | 3 | 4
Anorectal infection (Infections and infestations) | 3 | 4
Infections,other (Infections and infestations) | 2 | 5
Skin infection (Infections and infestations) | 2 | 4
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 45 | 20
back pain (Musculoskeletal and connective tissue disorders) | 3 | 4
Musculoskeletal disorder, other (Musculoskeletal and connective tissue disorders) | 5 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0
Skin and subcutaneous tissue disorder, other (Skin and subcutaneous tissue disorders) | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No